CLINICAL TRIAL: NCT04017130
Title: A Phase 1, Open-Label, Dose-Escalation, Multicenter Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of MT-0169 in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: A Study of MT-0169 in Participants With Relapsed or Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sparse/no patient enrollment
Sponsor: Molecular Templates, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: MT-0169-001; U1111-1224-6002 (Other: WHO); 2019-000931-24 (EudraCT Number)
Record Dates: First submitted 2019-07-10; First posted 2019-07-12 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Relapsed and/or Refractory Multiple Myeloma
Keywords: Drug therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Part 1: Dose Escalation (Experimental): Weekly Dosing Intravenous (IV) infusion of MT-0169 every 7 days: Days 1, 8, 15, and 22 in a 28-day treatment cycle.
  Every 2 Weeks IV infusion of MT-0169 every 14 days: Days 1 and 15 in a 28-day treatment cycle with escalating doses starting at the MTD/RP2D determined by the weekly dose escalation cohort.
  Patients will continue to receive treatment until progressive disease, unacceptable toxicity or withdraw from the study for other reasons. Decision to escalate/deescalate/stay on the same dose/discontinue MT-0169 will be based on number of DLTs per number of patients enrolled at each dose level as predetermined by the mTPI-2 statistical model. Subsequent doses will be determined by the frequency and severity of adverse events in previous cohorts. The investigator and sponsor review of available safety, PK, pharmacodynamics, and efficacy data in the previous cohorts will also be factored in the decision.
  Interventions: Drug: MT-0169

INTERVENTIONS:
Drug: MT-0169 — MT-0169 intravenous infusion.

SUMMARY:
This will be a Phase 1 Open-Label, dose escalation of MT-0169 (an Engineered toxin body (ETB) in patients with relapsed or refractory multiple myeloma. MT-0169 is an investigational drug that recognizes and binds to the CD38 receptor, which may be found on the surface of multiple myeloma cancer cells. It delivers a dose of a modified toxin that kills these cells.

DETAILED DESCRIPTION:
The drug being tested in this study is called MT-0169. The study will evaluate the safety, tolerability, preliminary efficacy, PK, pharmacodynamics, and immunogenicity of MT-0169 monotherapy in participants with RRMM.

The study will enroll up to 54 total participants.

The purpose of this study is to evaluate the safety and tolerability of MT-0169 in subjects with relapsed or refractory multiple myeloma (RRMM) and to estimate the maximum tolerated dose (MTD) or the recommended Phase 2 dose (RP2D).

MT-0169 will be given as an intravenous (IV) infusion over 60 minutes on the same day every week (i.e., days 1, 8, 15 and 22) or every 2 weeks (i.e., days 1 and 15) of each cycle. A cycle is defined as 28 days.

A subject may participate for the following three (3) periods:

Screening Period - up to 28 days before first dose of MT-0169 Treatment Period - active period where a subject will receive doses of MT-0169 over a 28-day treatment period Follow-up Period - up to 12 months after the last patient in the study to receive the last dose of MT-0169.

Participants can receive MT-0169 until the cancer worsens, side effects prevent further study treatment, or until the participant leaves the study for other reasons decided by the participant, the study doctor, or the sponsor of the study. After treatment has finished, participants will have a check-up of their disease status every 12 weeks.

This multi-center trial will be conducted in the United States. The overall duration of the study will vary for each participant because they will receive study treatment until unacceptable toxicity, withdrawal of consent, death, termination of the study by the sponsor, or fulfillment of another discontinuation criterion. Participants will be followed up for 30 days after the last dose of study drug for a follow-up assessment for any side effects. Participants will then be followed every 12 weeks to check for the status of their disease up to 12 months after the last subject on the trial has the last dose of study drug, or the sponsor discontinues the study, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria

1. Confirmed diagnosis of MM per revised IMWG diagnostic criteria
2. Patients with RRMM who have failed treatment with, are intolerant to, or are not candidates for available therapies that are known to confer clinical benefit
3. Must meet all of the following criteria for prior therapy:

   1. Must be refractory to ≥1 proteasome inhibitor (PI), ≥1 immunomodulatory drug (IMiD), and ≥1 steroid
   2. Must either have received ≥3 prior lines of therapy or ≥2 prior lines of therapy if 1 line included a combination of PI and IMiD (prior treatment with anti-CD38 therapy is permitted).
4. With measurable disease, defined as ≥1 of the following:

   1. Serum M-protein ≥500 mg/dL (≥5 g/L) on serum protein electrophoresis (SPEP).
   2. Urine M-protein ≥200 mg/24 h on urine protein electrophoresis (UPEP).
   3. Serum FLC assay result with an involved FLC level ≥10 mg/dL (≥100 mg/L) if serum FLC ratio is abnormal.
5. Patients with serum M-protein, urine M-protein, or involved immunoglobulin FLC not meeting the measurable disease criteria above will be eligible if they have ≥1 of the following:

   1. Bone marrow (BM) aspirate/biopsy with plasma cell percentage ≥30%
   2. PET imaging with ≥1 plasmacytoma lesion with a single diameter of ≥2cm.
6. With Eastern Cooperative Oncology Group (ECOG) performance score of 0 or 1.
7. With the following cardiovascular parameters:

   1. Left ventricular ejection fraction (LVEF) > 50% by echocardiogram or cardiac MRI.
   2. Cardiac troponin (high sensitivity or conventional) and NT-proBNP or BNP values within the institutional normal range
   3. QT interval corrected by the Fridericia method (QTcF) on screening electrocardiogram (ECG)[ QTcF of ≤450 millisecond (ms) in males or ≤470 ms in females]
8. Must meet the following clinical laboratory criteria at entry:

   1. Total bilirubin ≤1.5*the upper limit of the normal range (ULN), except for Gilbert's syndrome (direct bilirubin must be <2.0*ULN)
   2. Serum alanine aminotransferase (ALT), aspartate aminotransferase (AST) ≤2.5*ULN.
   3. Estimated glomerular filtration rate (eGFR) ≥30 (mL/min/1.73 square meter [m2]), using the modification of diet in renal disease (MDRD) equation
   4. Absolute neutrophil count (ANC) ≥1000 per cubic millimeter (/mm3) (≥1.0*109 per liter [/L]); ≥750/mm3 (≥0.75*109/L) may be acceptable for participants with >50% of plasma cells in BM
   5. Platelet count ≥75,000/ mm3 (≥75*109/L); ≥50,000/ mm3 (≥50*109/L) may be acceptable for participants with ≤ 50% of plasma cells in BM
   6. Hemoglobin ≥7.5 g/dL without transfusion within 7 days before the lab test.
   7. Serum albumin ≥2.5 g/dL.
9. Female patients who:

   1. are postmenopausal for at least 1 year prior to screening OR
   2. are surgically sterile OR
   3. If they are of childbearing potential, agree to practice 1 highly effective method of contraception and 1 additional effective barrier method at the same time from study entry through 30 days after the last dose of study drug OR
   4. agree to practice true abstinence if in line with the preferred, usual lifestyle [periodic abstinence (e.g., calendar, ovulation, symptothermal, postovulation methods), withdrawal, spermicides only, and lactational amenorrhea are not acceptable. Female and male condoms should not be used together]
10. Male patients, even if surgically sterilized (postvasectomy) who:

    1. Agree to practice effective barrier contraception during the entire study and through 90 days after last dose of study drug OR
    2. Agree to practice true abstinence if in line with the preferred, usual lifestyle [periodic abstinence (e.g., calendar, ovulation, symptothermal, postovulation methods), withdrawal, spermicides only, and lactational amenorrhea are not acceptable. Female and male condoms should not be used together]
11. Confirmed diagnosis of MM per IMWG diagnosis criteria:
12. RRMM, having failed treatment with, is intolerant to, or is determined not to be a candidate for available therapies considered SOC or are known to confer clinical benefit.
13. Must meet the following criteria for prior therapy:

    1. Refractory or intolerant to at least 1 proteasome inhibitor (PI) and at least 1 immunomodulatory drug (IMiD), and at least 1 steroid.
    2. Receipt of ≥3 prior lines of therapy, including a PI, an IMiD, and an anti-CD38 therapy such as daratumumab and isatuximab.
14. Measurable disease, defined as ≥1 of the following

    1. Serum M-protein ≥50 mg/dL (≥5 g/L) on SPEP.
    2. Urine M-protein ≥200 mg/24 hours on UPEP.
    3. Serum FLC assay result with and involved FLC level ≥10 mg/dL (≥100mg/L), provided the serum FLC ratio is abnormal.
15. Serum M-protein, urine M-protein or involved immunoglobulin FLC not meeting measurable disease criteria if they have extramedullary disease with either:

    1. Imaging showing at least 1 extramedullary lesion (except CNS listed below that has a single diameter of ≥2 cm, or
    2. Plasma cell leukemia.

Exclusion Criteria:

1. With polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy and skin changes (POEMS) syndrome, monoclonal gammopathy of unknown significance, smoldering myeloma, amyloidosis, Waldenström macroglobulinemia, or Immunoglobulin M (IgM) myeloma.
2. With sensory or motor neuropathy of NCI CTCAE V5 Grade ≥3.
3. Have received final dose of any of the following treatments/procedures within the following interval before the first dose of MT-0169:

   * Myeloma-specific therapy, including PIs and IMiDs: 14 days
   * Anti-CD38 (a) therapy: Isatuximab 90 days; daratumumab 60 days
   * Corticosteroid therapy for myeloma: 7 days
   * Radiation therapy for localized bone lesions: 14 days
   * Major surgery:30 days
   * Autologous stem cell transplant: 90 days
   * Investigational therapy: 30 days
4. Have received an allogeneic stem cell transplant or organ transplantation.
5. Have not recovered to Grade ≤1 or baseline, from adverse reactions to prior myeloma treatment or procedures (chemotherapy, immunotherapy, radiation therapy) excluding alopecia and Grade 2 neuropathy.
6. With clinical signs of central nervous system (CNS) involvement of MM.
7. With a history of myelodysplastic syndrome or another malignancy other than MM except for the following: any malignancy in complete remission for 3 years, adequately treated local basal cell or squamous cell carcinoma of the skin, cervical carcinoma in situ, superficial bladder cancer, or asymptomatic prostate cancer without known metastatic disease and not requiring therapy or requiring only hormonal therapy and with normal prostate-specific antigen level for ≥1 year before the start of study therapy.
8. With known or suspected light chain amyloidosis of any organ (amyloid on the BM biopsy without other evidence of amyloidosis is acceptable).
9. With any of the following cardiovascular conditions:

   1. Congestive heart failure (NYHA) class ≥II or cardiomyopathy, active ischemia, or any other uncontrolled cardiac condition or myocardial infarction or clinically significant arrhythmia requiring therapy including anticoagulants within the past 6 months or at screening (stable therapy for > 6 months is acceptable).
   2. Resting tachycardia (heart rate of > 100 bpm) at screening
   3. Clinically significant uncontrolled hypertension at screening
   4. Cardiac MRI at screening demonstrates evidence of amyloid cardiomyopathy or myocarditis
10. With a history of documented significant pleural or pericardial effusions of at least CTCAE Grade 3 within 3 months before the start of treatment. This will also exclude patients with:

    1. Pericarditis (any Grade)
    2. Non-malignant pleural effusion (Grade ≥2)
11. Patients with a history of noncardiogenic pulmonary edema associated with diffuse peripheral edema and history of intravascular hypovolemia associated with systemic antineoplastic therapy.
12. With chronic or active infection requiring systemic therapy, history of symptomatic viral infection that has not been fully cured. The following exceptions apply for those with positive serologies of HIV, HBV, or HCV:

    1. With HIV and an undetectable viral load and CD4+ T-cell (CD4+) counts ≥350 cells/mL may be allowed but patient must be taking appropriate opportunistic infection prophylaxis if clinically relevant
    2. With positive HBV serology may be allowed if undetectable viral load, receiving antiviral prophylaxis for potential HBV reactivation per institutional guidelines
    3. With positive HCV serology may be allowed if quantitative PCR for plasma HCV RNA is below the lower limit of detection. Concurrent antiviral HCV treatment per institutional guidelines is allowed.
13. Have received a live attenuated vaccine within 28 days of first dose of MT-0169.
14. With a history of CTCAE Grade 3 ≥ systemic inflammatory response syndrome (SIRS)/ cytokine release syndrome (CRS) reactions following infusion with any monoclonal antibodies (mAbs) or Chimeric Antigen Receptor (CAR) T therapy
15. With a chronic condition requiring systemic corticosteroids at >10 mg/day of prednisone or equivalent.
16. Are lactating and breastfeeding or have a positive serum pregnancy test during the screening period or patients of reproductive potential who are not employing an effective birth control
17. With a concurrent medical or psychiatric illness that would preclude study conduct and assessment including, but not limited to, uncontrolled medical conditions, active infection, risk of bleeding, diabetes mellitus, pulmonary disease, alcoholic liver disease, or primary biliary cirrhosis.
18. With known allergy or intolerance to any of the drugs used in the study or excipients in MT-0169
19. With a history of hypersensitivity or serious toxic reaction to kanamycin or another aminoglycoside.
20. Failed to recover to Grade ≤1 or baseline from adverse reactions to prior treatment or procedures (chemotherapy, immunotherapy, radiation therapy) excluding alopecia and stable Grade 2 neuropathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-02-05 (Actual); Primary Completion 2023-12-13 (Actual); Study Completion 2023-12-13 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) or recommended phase 2 dose (RP2D) | Up to 12 months
Number of participants with Treatment-emergent Adverse Events (TEAEs) | Up to 12 months
Number of participants with Dose-limiting Toxicities (DLTs) | Up to 12 months
Number of participants with Grade greater than or equal to (>=) 3 TEAEs according to NCI CTCAE 5.0 | Up to 12 months
Number of participants with Serious Adverse Events (SAEs) | Up to 12 months
Number of participants who discontinued MT-0169 due to TEAEs | Up to 12 months
Number of participants with treatment-related dose modifications | Up to 12 months
  Dose modifications include dose delays, dose interruptions, and dose reductions

SECONDARY OUTCOMES:
Cmax: maximum observed concentration for MT-0169 | Cycles 1 and 2, Day 1: pre-dose, and at multiple time points (up to 168 hours) post-dose (each cycle is 28 days)
Tmax: time to reach maximum observed concentration for MT-0169 | Cycles 1 and 2, Day 1: pre-dose, and at multiple time points (up to 168 hours) post-dose (each cycle is 28 days)
AUClast: Area Under the Concentration-time Curve From Time 0 to the time of the last quantifiable concentration for MT-0169 | Cycles 1 and 2, Day 1: pre-dose, and at multiple time points (up to 168 hours) post-dose (each cycle is 28 days)
Overall response rate (ORR) | Up to 12 months
  As defined by IMWG Uniform Response Criteria for RRMM patients.
Clinical Benefit Rate (CBR) for RRMM patients | Up to 12 months
  Percentage of participants who achieved PR or better during study as defined by IMWG Uniform Response Criteria and ORR in patients with RRNHL as defined by the Lugano classification for lymphoma.
Progression-free Survival (PFS) for RRMM patients | From the date of first dose until the date of progressive disease (PD)
  Determined by IMWG criteria
Proportion of RRMM participants who achieved MR (minimal response) | Up to 12 months
  MR is defined as the percentage of participants who achieved 25% tumor reduction.
Duration of Response (DOR) | Date of the dose administration until death due to any cause (up to 12 months)
  Time from the date of the first documentation of response to the date of the first documented PD.
Number of participants with Anti-drug Antibodies following administration of MT-0169 | Up to 12 months
Overall survival (OS) | From date of the dose administration until death due to any cause (up to 12 months)
Time to Response (TTR) | From the date of the first dose of the study treatment to the date of the first documentation of response (up to 12 months)
Percentage of participants with RRMM who achieved Complete Response (CR) or Very Good Partial Response (VGPR) | Up to 12 months

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - University of Southern California, Los Angeles, California
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Miami University, Miami, Florida
  - Northside Hospital, Atlanta, Georgia
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - The Ohio State University, Columbus, Ohio
  - Vanderbilt University Medical Center- Ingram Cancer Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No